CLINICAL TRIAL: NCT03080441
Title: Minimization of Intradialytic Hypotension Using Cardiography-Guided Intervention
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Nimedical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIM01
Record Dates: First submitted 2017-02-08; First posted 2017-03-15 (Actual); Last update posted 2017-03-15 (Actual); Status verified 2017-03

CONDITIONS: Intradialytic Hypotension
MeSH Terms: interventions — Stockings, Compression; Midodrine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Phase 1 Group 1 (Experimental): pressure stockings worn during dialysis treatment
  Interventions: Device: pressure stockings
- Phase 1 Group 2 (Experimental): Midodrine before dialysis treatment
  Interventions: Drug: Midodrine
- Phase 1 Group 3 (Experimental): pressure stocking and Midodrine
  Interventions: Other: pressure stockings and midodrine

INTERVENTIONS:
Device: pressure stockings — pressure stockings worn during dialysis throughout treatment period
  Arms: Phase 1 Group 1
Drug: Midodrine — administered Midodrine before each dialysis treatment during treatment period based on PI's judgement. Including consideration of blood pressure.
  Arms: Phase 1 Group 2
Other: pressure stockings and midodrine — combination of Midodrine and pressure stocking before each dialysis treatment throughout treatment period
  Arms: Phase 1 Group 3

SUMMARY:
This is a research study to test the application of FDA-approved, non-invasive device (NICaS) that measure the performance of your heart during HD treatment.

DETAILED DESCRIPTION:
The incidence of intradialytic hypotension (IDH) events, reported to occur in 15% to 50% of hemodialysis (HD) treatments, is still high despite major technical advances in HD technology. By definition, excessive reduction in intravascular volume by ultrafiltration and limited vascular refilling from tissues into the vascular space is the cause of IDH. Chronic HD patients exhibit a high prevalence of peripheral vascular and cardiac abnormalities. Specifically, hemodynamic instability during HD can occur due to insufficient reduction in venous unstressed volume, poor diastolic filling under reduced atrial pressures associated with diastolic dysfunction, altered cardiac contractility, and impaired vascular reactivity. An IDH event can lead to myocardial cerebral and other organ ischemia. Long- and short-term adverse outcomes have been associated with IDH, a common HD complication and significant cause of morbidity.

Recent pilot studies suggest that in IDH-prone subjects, measurements of hemodynamic variables during HD can be used to categorize the hemodynamic response into three subgroups: cardiac power index (CPI) reduction with stable total peripheral resistance (TPR), TPR reduction with stable CPI, and reduction in TPR and CPI groups. It is hypothesized that targeted intervention for each subgroup can reduce IDH.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* Have been on maintenance hemodialysis at the facility for at least six months
* Have not had un-excused missed treatments for six months
* Is symptomatic to HD treatments
* Males and non-pregnant/non-nursing females, as confirmed via urine pregnancy testing of women of child bearing potential

Exclusion Criteria:

* Patient refusal
* Currently on Midodrine at the start of the Phase 1, Observation period
* Any known contraindications to Midodrine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2016-11-11 (Actual); Primary Completion 2017-04-01 (Estimated); Study Completion 2017-05-01 (Estimated)

PRIMARY OUTCOMES:
Hypotension | 6 weeks
  Post dialysis BP measured in mm/Hg
Weight | 6 weeks
  Post dialysis weight measure in kg
Cardiac Index | 1 week
  Cardiac Index results from NICaS results vs Echocardiogram results measured in L/min/m2

IPD SHARING:
Plan to Share IPD: No
There is no current plan to share IPD with other researchers